CLINICAL TRIAL: NCT03823014
Title: Use of an External Erectile Device in Transgender Man Following Phalloplasty
Acronym: ProstHEsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Boskey, Researcher, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00029965
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Transsexualism; Surgery; Sex Behavior; Erectile Dysfunction
Keywords: transgender; transmasculine; ftm; phalloplasty; penile prosthesis
MeSH Terms: conditions — Transsexualism; Sexual Behavior; Erectile Dysfunction; Meckel Syndrome, Type 5

STUDY DESIGN:
Intervention Model Description: Pilot study to determine feasibility of device use for supportive care of transgender patients with erectile concerns post phalloplasty. Device is currently available in market.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- External Erectile Prosthesis (Experimental): Study participants will be recruited as couples (transgender man + sexual partner.) Couples will use an external erectile prosthesis (Elator) over the course of 1 month and keep track of their experiences. 20 men and their partners will be enrolled.
  Interventions: Device: Elator

INTERVENTIONS:
Device: Elator — Measurement for device, use of device
  Other Names: Erector

SUMMARY:
The purpose of this study is to test whether an external erectile prosthesis (The Elator™) is a feasible alternative to internal erectile prostheses for transgender men who have undergone a phalloplasty with glansplasty and wish to use their neophallus for sexual penetration. The Elator™ was initially developed for men experiencing erectile dysfunction after prostate cancer. The device consists of two silicone rings connected by a pair of plastic coated rigid metal rods. One ring goes at the base of the penis. The other ring is connected to the rods. This ring is placed behind the glans, and then the rods are connected to the base ring to stretch and provide rigidity to the phallus.

DETAILED DESCRIPTION:
There are approximately 1.4 million transgender adults in the United States. Approximately half are transgender men, individuals who have a male gender identity but were assigned female at birth. A national survey of transgender adults found more than half of transgender men have had, or may want, gender affirmation surgery in the form of phalloplasty - the surgical creation of a penis and scrotum. The neophallus created in this manner can be used for standing urination but not for penetrative sex, due to the lack of erectile structures.

Research suggests that one factor limiting interest in phalloplasty is the lack of reliable, durable, and desirable erectile devices. Internal prostheses are the primary method used to attain penile rigidity after phalloplasty. However, these devices carry a significant risk of mechanical failure and other adverse events. The high failure and complication rates associated with internal erectile prostheses demonstrate a need for alternative options for transgender men after phalloplasty. One such option consists of an external erectile prosthesis or support. The Elator™ consists of two silicone rings connected by a pair of plastic coated rigid metal rods. Use of such an external device may be preferable for men who do not wish to undergo additional surgery after phalloplasty, and/or those who have had problems with internal prostheses.

Word of mouth suggests that a number of transgender men have experimented with these devices after phalloplasty, but to date no study has tested the safety and function of external erectile prostheses in this population. Currently, the FDA exempts most external penile rigidity devices from pre-market notification and review. As such, safety and efficacy testing is not required prior to public marketing. However, before medical professionals can feel comfortable recommending these devices to their patients, such testing is clearly indicated.

The proposed pilot study will test whether an external erectile prosthesis (The Elator™) is a feasible alternative to internal erectile prostheses for transgender men after phalloplasty. This study will recruit twenty men who have had a phalloplasty greater than one year prior to the study date, have protective sensation to the tip of their phallus, have a current sexual partner with whom they would like to explore sexual penetration using the neophallus, and who do not currently have an internal erectile prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Primary study subject must have had a phalloplasty with glansplasty a minimum of 1 year before enrollment and must have protective sensation to the tip of the phallus
* Primary study subject must be in a relationship in which they are having, or would like to have, penetrative sex with their partner. Partner must also be interested in having penetrative sex with primary subject.
* Both primary study subject and partner must have (individual) e-mail addresses and access to the Internet to complete surveys
* Primary study subject must be willing to be contacted by postal mail, in order to receive the device
* Both subjects must be willing to receive e-mails

Exclusion Criteria:

* Either subject or partner does not speak English
* Primary subject has an internal erectile prosthesis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender men and their sexual partners (no gender/sex requirement)
Enrollment: 15 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Sexual Experience Scale | Baseline and at study completion (~1.5 months)
  Brief measure of quality of most recent sexual experience
Change in Relationship Satisfaction Subscale | Baseline and at study completion (~1.5 months)
  Measure of overall relationship satisfaction with romantic partner
Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) | The intervention period of 4 weeks, assessed at study completion
  Validated measure of satisfaction with erectile dysfunction treatment

SECONDARY OUTCOMES:
Qualitative Device Feedback | The intervention period of 4 weeks, assessed at study completion
  Interview with men and their partners about the experience of using the device (optional)

CONTACTS AND LOCATIONS:
Locations (1):
- Participation in this study is from participants home., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No